CLINICAL TRIAL: NCT06507137
Title: Fractal-based Gait Training in Older Adults: Implications to Motor Control and Neuroplasticity
Brief Title: Fractal-based Gait Training in Older Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: FRACTRAIN-1378/24
Record Dates: First submitted 2024-06-19; First posted 2024-07-18 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Healthy Aging
Keywords: Gait Rehabilitation; Aging; Neuroscience; Falls Prevention; Dynamical Systems
MeSH Terms: interventions — Fractals

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fractal (Experimental)
  Interventions: Other: Fractal
- Isochronous (Experimental)
  Interventions: Other: Isochronous
- Control (Experimental)
  Interventions: Other: Control

INTERVENTIONS:
Other: Fractal — Walking in a treadmill while synchronizing their steps with fractal external visual cues
  Arms: Fractal
Other: Isochronous — Walking in a treadmill while synchronizing their steps with isochronous external visual cues
  Arms: Isochronous
Other: Control — Walking in a treadmill
  Arms: Control

SUMMARY:
The purpose of the study is to investigate the influence of walking with external visual cues on brain adaptations.

ELIGIBILITY:
Exclusion Criteria:

* Neurologic conditions;
* Lower limb disabilities or disease;
* Not able to provide informed consent;
* Unable to walk unassisted for 10-minutes continuously;
* Score below 24 in the Mini-Mental State Examination (MMSE);
* Have a history of falls in the prior six months;
* Have an implanted device (e.g., pacemakers);
* Medication advised against the application of Transcranial Magnetic Stimulation.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Fractal scaling exponent (α) changes from baseline (PRE to POS, PRE to FUP, POS to FUP) both within and between Fractal, Isochronous and Control groups. | PRE (baseline), POS (4 weeks after), FUP (8 weeks after)
  The fractal scaling exponent quantifies the complexity of a physiological signal and detects the presence of statistical persistence in a given time series. This parameter is calculated using Detrended Fluctuation Analysis (DFA) from each time series (stride time and stride length).

SECONDARY OUTCOMES:
Corticospinal excitability (CSE) changes from baseline (PRE to POS, PRE to FUP, POS to FUP) both within and between Fractal, Isochronous and Control groups. | PRE (baseline), POS (4 weeks after), FUP (8 weeks after)
  CSE is a parameter extracted through the application of Transcranial Magnetic Stimulation (TMS). This parameter provides information regarding the level of excitability of the corticospinal tract.
Short-Interval Intracortical Inhibition (SICI) changes from baseline (PRE to POS, PRE to FUP, POS to FUP) both within and between Fractal, Isochronous and Control groups. | PRE (baseline), POS (4 weeks after), FUP (8 weeks after)
  SICI is a parameter extracted through the application of Transcranial Magnetic Stimulation (TMS). This parameter provides information regarding the level of inhibition of the motor cortex.
Intracortical Facilitation (ICF) changes from baseline (PRE to POS, PRE to FUP, POS to FUP) both within and between Fractal, Isochronous and Control groups. | PRE (baseline), POS (4 weeks after), FUP (8 weeks after)
  ICF is a parameter extracted through the application of Transcranial Magnetic Stimulation (TMS). This parameter provides information regarding the level of facilitation of the motor cortex.
Ankle, Knee and Hip joints range of motion's changes from baseline (PRE to POS, PRE to FUP, POS to FUP) both within and between Fractal, Isochronous and Control groups during a gait cycle | PRE (baseline), POS (4 weeks after), FUP (8 weeks after)
  Joint range of motion is measured through a motion capture system and quantifies the excursion of the joint during the gait task in degrees (º).
Ankle, Knee and Hip joints maximum value changes from baseline (PRE to POS, PRE to FUP, POS to FUP) both within and between Fractal, Isochronous and Control groups during a gait cycle | PRE (baseline), POS (4 weeks after), FUP (8 weeks after)
  Joint maximum value is measured through a motion capture system and quantifies the maximum joint flexion during the gait task in degrees (º). This measure will be used to calculate joint range of motion (outcome 2).
Ankle, Knee and Hip joints minimum value changes from baseline (PRE to POS, PRE to FUP, POS to FUP) both within and between Fractal, Isochronous and Control groups during a gait cycle | PRE (baseline), POS (4 weeks after), FUP (8 weeks after)
  Joint minimum value is measured through a motion capture system and quantifies the minimum joint flexion during the gait task in degrees (º). This measure will be used to calculate joint range of motion (outcome 2).
Ankle, Knee and Hip joints angles during initial contact changes from baseline (PRE to POS, PRE to FUP, POS to FUP) both within and between Fractal, Isochronous and Control groups during a gait cycle | PRE (baseline), POS (4 weeks after), FUP (8 weeks after)
  Joint angle during initial contact is measured through a motion capture system and quantifies the angle of the respective joint at the moment the heel touches the ground during a gait cycle (heel strike) in degrees (º).
Ankle, Knee and Hip joints angles during peak ground reaction force changes from baseline (PRE to POS, PRE to FUP, POS to FUP) both within and between Fractal, Isochronous and Control groups during a gait cycle | PRE (baseline), POS (4 weeks after), FUP (8 weeks after)
Coefficient of variation (CV) changes from baseline (PRE to POS, PRE to FUP, POS to FUP) both within and between Fractal, Isochronous and Control groups. | PRE (baseline), POS (4 weeks after), FUP (8 weeks after)
  CV is a common linear measure that translates the amount of variability within the signal and is calculated through the standard deviation normalised to the mean from each time series (stride time and stride length).
Electromyography co-contraction changes from baseline (PRE to POS, PRE to FUP, POS to FUP) both within and between Fractal, Isochronous and Control groups. | PRE (baseline), POS (4 weeks after), FUP (8 weeks after)
  Co-contraction is the simultaneous activation of the agonist and antagonist muscles during a task. This parameter It is an important mechanism of the central nervous system to regulate joint stability and provide movement accuracy.

CONTACTS AND LOCATIONS:
Locations (1):
- Egas Moniz School of Health and Science, Almada, Monte de Caparica, Portugal

IPD SHARING:
Plan to Share IPD: No